CLINICAL TRIAL: NCT04737993
Title: Pulsed Radiofrequency of Suprascapular Nerve and Shoulder Joint for Chronic Shoulder Pain: A Randomized Blind Active -Controlled Study
Brief Title: Pulsed Radiofrequency of Suprascapular Nerve and Shoulder Joint for Chronic Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Satasairaala (Other)
Responsible Party: Principal Investigator, Hannu heikkilä, Head of unit for physical medicine and rehabilitation, Satasairaala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1184/13.01/2018
Record Dates: First submitted 2020-12-16; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Chronic Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- prf shoulder joint (Active Comparator): pulsed rf stimulation of joint capsel and prf stimlation of subscapular nerve
  Interventions: Drug: licocain; Other: pulsed radiofrequency stimulation
- prf subscapular nerve (Active Comparator): pulsed RF stimulation of subscapular nerve
  Interventions: Drug: licocain; Other: pulsed radiofrequency stimulation
- subscapular nerve block (Active Comparator): lidocain injection of subscapular nerve
  Interventions: Drug: licocain

INTERVENTIONS:
Drug: licocain — pulsed radiofrequency stimulation
  Other Names: radiofrequency stimulation
Other: pulsed radiofrequency stimulation — pulsed radiofrequency stimulation of joint capsel
  Arms: prf shoulder joint; prf subscapular nerve

SUMMARY:
Background: The suprascapular nerve block is frequently used to treat chronic shoulder pain. The nerve blockade provides probably only a short-term relief, and more compelling approaches have been investigated. Pulsed radiofrequency stimulation of suprascapular nerve has been reported as safe and reliable method for pain treatment. However, formal efficacy study for pRF stimulation of the shoulder joint has not been published. Evidence-based validation of a new method is necessary for both scholastic and practical purposes.

Methods: This study is a randomized active controlled blind trial. Lidocaine injections alone and pRF stimulation with two different combinations will be performed. Participants will be followed during 6 months, and subjective and objective outcome variables will be recorded. Patients are randomly allocated for suprascapular nerve block (n=50), for suprascapular nerve pRF stimulation (n=50) or for both suprascapular nerve blocks and humeroscapular joint pRF stimulation (n=50). All patients will receive standardized physical therapy at the unit of physical medicine and rehabilitation.

Results: Pulsed radiofrequency is thought to be a non-neurolytic neuromodulation method with some effectiveness in relieving of both experimental and clinical neuropathic pain. Our earlier results suggest additional therapeutic benefit obtained when pRF was performed in addition to physiotherapy (TAU). In a review, Chan et al. (2016) concluded that SSNB treatment could be more effective in treating pain in patients with longstanding rheumatoid arthritis when compared to intra-articular injection of corticosteroid. Also short-term pain reduction occurred in patients with chronic rotator cuff lesions. With regard to adhesive capsulitis, SSNB treatment showed a greater effect in relieving pain but on functional outcome, the results were inconclusive.

Discussion: In summary, this study investigate effects of pRF for patients with chronic shoulder pain from arthritis, frozen shoulder and/or degenerative shoulder disease. PRF can be performed in an outpatient department and provides the clinician with an alternative or additional approach to oral drug treatment and intra-articular injection. Further, it may prove to be a useful treatment for patients who are unfit or unwilling to consider surgical intervention.

DETAILED DESCRIPTION:
Introduction After spinal and knee pain, shoulder pain is estimated to be the third most common type of musculoskeletal pain, causing considerable psychosocial impact if progressing to the chronic phase. While majority of patients with shoulder pain recover within few months, over 40% of patients have persisting symptoms after 12 months. Establishing a treatment strategy for shoulder pain can be challenging, as the effectiveness of many treatment options is unclear. Non-surgical strategies are preferred in the first-line management, with physiotherapy being of the treatment of choice in the majority of cases. Physiotherapy, pain medication and corticosteroid injections (CSI) are used but the effectiveness of these interventions may be insufficient. Corticosteroid injections are often used in treatment of shoulder pain, though there is no clear evidence of long-term benefit. It has been reported that CSI might lead to adverse events such as tendon degeneration, cutaneous atrophy or infection. In addition, CSI can cause systemic side effects including changes in the hypothalamic-pituitary-adrenal axis function and elevated blood glucose levels. Therefore, safer pain management options with more long-lasting pain relief are sought. The suprascapular nerve derives from the ventral rami of cervical spinal nerves C4, C5, and C6 and arises from the upper trunk of the brachial plexus, contributes approximately 70% of the sensory innervation to the shoulder joint. Suprascapular nerve blocks have been used to manage acute and chronic shoulder pain, although the efficacy of treatment alters in different studies and when compared to other treatment options. The short duration of action of local anesthetics raises the question of their efficacy in the management of chronic shoulder conditions. In addition to SSNB, pulsed radiofrequency stimulation (pRF) has also been researched for its potentially greater and longer-lasting outcomes when comparing to local anesthetics. There has been limited numbers of reviews specifically investigating the usefulness of SSNB for the treatment of chronic shoulder pain. Liu et al. concluded in their review pRF treatment to result in good efficiency in shoulder patients with no significant complications reported. The pain relief could last several months. Only few case reports have been made on pRF treatment of the glenohumeral joint. Considering the adverse effects of corticosteroids, SSNB with local anesthetics could be regarded as a potential alternative for pain relief in patients who have adhesive capsulitis. Our earlier results suggested additional therapeutic benefit obtained when pRF for both suprascapular nerve and shoulder joint was performed in addition to physiotherapy.

The aim of this study was to compare whether pRF treatment of both glenohumeral joint and suprascapular nerve provided additional clinical benefits compared to suprascapular nerve block or pRF treatment of suprascapular nerve only. The rehabilitation included also individual functional training and treatment as recommended by the national task group.

Method This randomized controlled trial will follow the Consolidated Standards of Reporting Trials Statement; it will be performed at Central Hospital in Satakunta, Pori, Finland. The study has been approved by the local Research Ethics Committee (SS/1184/13.01/2018). The sample size estimate was obtained to detect differences between the treatment groups in relation to the primary outcome of the study after the intervention. Kukkonen's et al. study estimated the clinically important minimal difference in CM score in 10.4 points in patients with rotator cuff rupture after 3 months of surgical treatment by the arthroscopic method. The estimated sample size of 45 patients per group, total of 135patients, would reach 90% power to detect a 10.4 difference between the groups in the SPADI instrument follow-up score with a standard deviation of up to 15 points with a significance level of 5% using a t-Student test. Predicting a loss of around 10% at 6 months follow-up, we aim to recruit 50 patients per group. The placebo response is usually estimated as high as 30%. Using calculation of difference between proportions, the sample size was estimated as 50 patients total. Randomization 1:1:1 is performed. Patients will be consecutively allocated to one of three proposed treatment methods. The software R was used to generate a randomization list, considering 150 patients included in the study and the same probability of allocation for methods of pain treatment intervention. Patients with shoulder pain > 3 months duration, clinical and imaging confirmation of adhesive capsulitis, tendinosis, arthritis, rotator cuff or capsular tears are eligible for participation. Failure of conservative medical therapy is documented. Exclusion criteria comprised refusal to participate, extrinsic source of shoulder pain (e.g., cervical radiculopathy) and pain related to bony fracture. All patients are at first evaluated by specialist in physical medicine and rehabilitation who use ultrasound and clinical examination to estimate shoulder function. Patients who have more specific shoulder dysfunction based on subjective symptoms and clinical evaluation are asked to participate this intervention study. Of totally around 300 consecutive patients who receive pRF on the suprascapular nerve and shoulder joint, 150 consecutive patients are estimated voluntarily participate the study. Primary outcomes, such as Shoulder Pain and Disability Index ,15D self-administered measure of health-related quality of life and working ability are measured. This study is also part of the quality register study of the unit. Our standardized patient surveys cover demographic data, level of education, work status and future outlook, pain intensity, psychological factors, measurements of activity/participation and health-related quality of life (MPI, HAD SF-36, EQ-5D,CPAQ;Tampa,ISI). Those patients, who report no pain relief at 2-month follow-up and are dissatisfied, have an option to undergo pRF procedure any time after the first follow-up visit. Patients are able to dropout from the study any time. The randomization will be carried out by assisting nurse and delivered in sealed envelopes marked SSPS "subscapularis" (suprascapular nerve block), " pRF suprascapular" (pRF stimulation of suprascapular nerve) or "suprascapualar + joint" (pRF stimulation both suprascapular nerve and shoulder joint). Patient will be blinded. Two operators to minimize individual technical differences perform all procedures. Physician who did not treat the patient primarily and did not know which treatment patient received will conduct follow up estimation (pretreatment, 10 and 30 weeks after intervention). The groups will be compared according to the presence of categorical clinical outcomes by Chi-square or Fisher's exact tests, depending on the distribution observed after data collection. The analyzes will be performed with the aid of the SPSS program, considering a significance level of 5%. Demographic variables will be compared using a t-test or chi-squared test for continuous and categorical variables, respectively. Repeated measures ANOVA will be utilized for the primary outcome of Pain NRS and the secondary outcomes of the SPADI and AROM. Planned contrasts examining the linear trend effect of each group's scores over time were also included in the analysis. For the HRQoL scale, paired-sample t-tests will be conducted to compare groups, at each time.

Interventions All patients will be offered conservative treatment including pharmacotherapy (opioid analgesics, NSAIDs, paracetamol, adjuvant medication) and physiotherapy. Physiotherapy program based on manual therapy intervention focus on increasing function and pain control. Physical training is largely based on specific movements supervised by qualified physiotherapists. The emphasis is on individual training program, and on learning a functional use of the arm. PRF treatment and nerve block will be performed under ultrasound guidance. First, the suprascapular notch is identified using ultrasound with the patient in the sitting position, shoulders relaxed and forearms placed on the thighs. The puncture site is located on the line dividing the upper-outer quadrant of the scapula approximately 2.5 cm from the top. Following the puncture, an isolated radiofrequency 23-G 60 mm needle with a 5 mm active tip (Top Neuropole needle XE 60 mm 23G) is introduced perpendicularly to the skin in all planes. Selective stimulation of motor fibers (50 Hz) commenced after the needle tip had penetrated into the suprascapular notch. Motoric response or paresthesia at a voltage between 0.3 and 0.5 V is sought.

Envelopes marked SSPS "supraspinatus" will result in injection of 1 ml Lidocaine (10%) and "pRF suprascapularis" or "suprascapualris+joint" result in pRF stimulation, a 4-minute cycle of pRF with STP (Sluijter Teixeira Pulsed Poisson) program (TOP Lesion Generator TLG-10, Equip Medikey BV, The Netherlands) will be performed. One ml Lidocaine (10%) will be injected at the end of therapy since irritation of nerve fibers by the electrical field (without thermolesion) has been described as occurring frequently. Shoulder joint RF stimulation procedure use posterior approach. The sulcus between the head of the humerus and acromion is identified by ultrasound. The needle is inserted 2-3cm inferior and medial to the posterolateral corner of the acromion and directed anteriorly towards the coracoid process. An isolated radiofrequency 23-G 60 mm needle with a 5 mm active tip (Top Neuropole needle XE 60 mm 23G) will be introduced perpendicularly to the skin in all planes completely into the joint. First, 0,1-0,2 ml Lidocaine (10%) will be injected after puncture of skin and after pRF treatment 0,8 ml in the shoulder joint. Joint capsule stimulation, a 4 minute cycle of pRF with STP program is performed. Pain VAS, glenohumeral joint active range of motion and any complications will be recorded before discharge. The patients receive contact details of an available nurse prior to discharge. Next week after the RF-stimulation, we recommend restart of physiotherapy intervention focused on increasing function and pain control. Average rehabilitation time is calculated to be three months and on average patients have six consultations (1-12) in 6 months.

MEASUREMENTS Prior to the first MD appointment, participants are asked to compleat questionnaire. At the first appointment, using standardized clinical data forms; MD record the history of the participant's shoulder problem and clinical examination findings. In addition to active and passive ranges of motion, Visual Analogue Scale (VAS) and Shoulder Pain and Disability Index (SPADI), are recorded to assess shoulder function. The SPADI is a patient administered questionnaire consisting of 13 items divided into two subscales: pain (5 questions) and disability (8 questions). The pain and disability subscales are scored separately and then calculated into a total SPADI score, with higher scores demonstrating increased pain and disability. We also included 15D self-administered measure of health-related quality of life (HRQoL). 15D is a generic, comprehensive, 15-dimensional, standardized, self-administered measure of health-related quality of life (HRQoL) and it can be used as a profile and single index score measure. The single index score (15D score) on a 0-1 scale, representing the overall HRQoL, is calculated. Participants will be followed during 6 months, and subjective and objective outcome variables will be recorded for primary outcome instruments at 2 and 6 months and secondary outcome instruments at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

shoulder joint pain >3 moths

Exclusion Criteria:

Other ethiology as cervical root leasion or cancer.-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
SPADI change is being assessed | 0, 2, 6 months
  Shoulder Pain and Disability Index change from baseline is being assessed at 2 and 6 months . Disability, pain and total scores 0-100% when 100 is worst.
Active maximal shoulder adduction movement change is being assessed | 0,2,6 months
  Active shoulder joint adduction min 0- max 180. Change from baseline is being assessed at 2 and 6 months
Active maximal shoulder flexion movement change is being assessed | 0,2,6 months
  Active Shoulder joint flexion min 0 -max 180. Change from baseline is being assessed at 2 and 6 months

SECONDARY OUTCOMES:
HQoL 15 d change is being assessed | 0,6 months
  measure of health-related quality of life 15 items. Change from baseline is being assessed at 6 months. Questionnaire result in index, Minimum 0 and maximum1.
EQ5D change is being aseessed | 0, 6 months
  measure of health-related quality of life. Change from baseline is being assessed at 6 months. Questionnaire result in index, Minimum 0 and maximum1.

CONTACTS AND LOCATIONS:
Overall Officials: hannu v heikkilä, Study Director — Satasairaala
Locations (1):
- dep of physical medicine and rehabilitation Satasairaala, Pori, Finland

REFERENCES:
- [Background] Krismer M, van Tulder M; Low Back Pain Group of the Bone and Joint Health Strategies for Europe Project. Strategies for prevention and management of musculoskeletal conditions. Low back pain (non-specific). Best Pract Res Clin Rheumatol. 2007 Feb;21(1):77-91. doi: 10.1016/j.berh.2006.08.004. PMID 17350545
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Jensen I, Harms-Ringdahl K. Strategies for prevention and management of musculoskeletal conditions. Neck pain. Best Pract Res Clin Rheumatol. 2007 Feb;21(1):93-108. doi: 10.1016/j.berh.2006.10.003. PMID 17350546
- [Background] Linsell L, Dawson J, Zondervan K, Rose P, Randall T, Fitzpatrick R, Carr A. Prevalence and incidence of adults consulting for shoulder conditions in UK primary care; patterns of diagnosis and referral. Rheumatology (Oxford). 2006 Feb;45(2):215-21. doi: 10.1093/rheumatology/kei139. Epub 2005 Nov 1. PMID 16263781
- [Background] Silverstein BA, Viikari-Juntura E, Fan ZJ, Bonauto DK, Bao S, Smith C. Natural course of nontraumatic rotator cuff tendinitis and shoulder symptoms in a working population. Scand J Work Environ Health. 2006 Apr;32(2):99-108. doi: 10.5271/sjweh.985. PMID 16680380
- [Background] Coghlan JA, Buchbinder R, Green S, Johnston RV, Bell SN. Surgery for rotator cuff disease. Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD005619. doi: 10.1002/14651858.CD005619.pub2. PMID 18254085
- [Background] Saltychev M, Aarimaa V, Virolainen P, Laimi K. Conservative treatment or surgery for shoulder impingement: systematic review and meta-analysis. Disabil Rehabil. 2015;37(1):1-8. doi: 10.3109/09638288.2014.907364. Epub 2014 Apr 2. PMID 24694286
- [Background] Saltychev M, Virolainen P, Laimi K. Conservative treatment or surgery for shoulder impingement: updated meta-analysis. Disabil Rehabil. 2020 Jun;42(11):1634-1635. doi: 10.1080/09638288.2019.1622796. Epub 2019 May 30. No abstract available. PMID 31144999
- [Background] van der Windt DA, Koes BW, de Jong BA, Bouter LM. Shoulder disorders in general practice: incidence, patient characteristics, and management. Ann Rheum Dis. 1995 Dec;54(12):959-64. doi: 10.1136/ard.54.12.959. PMID 8546527
- [Background] Cook T, Minns Lowe C, Maybury M, Lewis JS. Are corticosteroid injections more beneficial than anaesthetic injections alone in the management of rotator cuff-related shoulder pain? A systematic review. Br J Sports Med. 2018 Apr;52(8):497-504. doi: 10.1136/bjsports-2016-097444. Epub 2018 Jan 5. PMID 29305377
- [Background] Buchbinder R, Green S, Youd JM. Corticosteroid injections for shoulder pain. Cochrane Database Syst Rev. 2003;2003(1):CD004016. doi: 10.1002/14651858.CD004016. PMID 12535501
- [Background] Habib GS, Saliba W, Nashashibi M. Local effects of intra-articular corticosteroids. Clin Rheumatol. 2010 Apr;29(4):347-56. doi: 10.1007/s10067-009-1357-y. Epub 2010 Jan 26. PMID 20101428
- [Background] Habib GS. Systemic effects of intra-articular corticosteroids. Clin Rheumatol. 2009 Jul;28(7):749-56. doi: 10.1007/s10067-009-1135-x. Epub 2009 Feb 28. PMID 19252817
- [Background] Muto T, Kokubu T, Mifune Y, Inui A, Harada Y, Yoshifumi, Takase F, Kuroda R, Kurosaka M. Temporary inductions of matrix metalloprotease-3 (MMP-3) expression and cell apoptosis are associated with tendon degeneration or rupture after corticosteroid injection. J Orthop Res. 2014 Oct;32(10):1297-304. doi: 10.1002/jor.22681. Epub 2014 Jul 2. PMID 24985902
- [Background] Nichols AW. Complications associated with the use of corticosteroids in the treatment of athletic injuries. Clin J Sport Med. 2005 Sep;15(5):370-5. doi: 10.1097/01.jsm.0000179233.17885.18. PMID 16162982
- [Background] Vorster W, Lange CP, Briet RJ, Labuschagne BC, du Toit DF, Muller CJ, de Beer JF. The sensory branch distribution of the suprascapular nerve: an anatomic study. J Shoulder Elbow Surg. 2008 May-Jun;17(3):500-2. doi: 10.1016/j.jse.2007.10.008. Epub 2008 Feb 11. PMID 18262803
- [Background] Dean BJ, Gwilym SE, Carr AJ. Why does my shoulder hurt? A review of the neuroanatomical and biochemical basis of shoulder pain. Br J Sports Med. 2013 Nov;47(17):1095-104. doi: 10.1136/bjsports-2012-091492. Epub 2013 Feb 21. PMID 23429268
- [Background] Borstad J, Woeste C. The role of sensitization in musculoskeletal shoulder pain. Braz J Phys Ther. 2015 Jul-Aug;19(4):251-7. doi: 10.1590/bjpt-rbf.2014.0100. Epub 2015 Aug 7. PMID 26443971
- [Background] Fernandes MR, Barbosa MA, Sousa AL, Ramos GC. Suprascapular nerve block: important procedure in clinical practice. Rev Bras Anestesiol. 2012 Jan-Feb;62(1):96-104. doi: 10.1016/S0034-7094(12)70108-3. PMID 22248771
- [Background] Chan CW, Peng PW. Suprascapular nerve block: a narrative review. Reg Anesth Pain Med. 2011 Jul-Aug;36(4):358-73. doi: 10.1097/AAP.0b013e3182204ec0. PMID 21654552
- [Background] Chang KV, Hung CY, Wu WT, Han DS, Yang RS, Lin CP. Comparison of the Effectiveness of Suprascapular Nerve Block With Physical Therapy, Placebo, and Intra-Articular Injection in Management of Chronic Shoulder Pain: A Meta-Analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2016 Aug;97(8):1366-80. doi: 10.1016/j.apmr.2015.11.009. Epub 2015 Dec 14. PMID 26701762
- [Background] Liu A, Zhang W, Sun M, Ma C, Yan S. Evidence-based Status of Pulsed Radiofrequency Treatment for Patients with Shoulder Pain: A Systematic Review of Randomized Controlled Trials. Pain Pract. 2016 Apr;16(4):518-25. doi: 10.1111/papr.12310. Epub 2015 May 19. PMID 25990576
- [Background] Ozyuvaci E, Akyol O, Acikgoz A, Leblebici H. Intraarticular pulsed mode radiofrequency lesioning of glenohumeral joint in chronic shoulder pain: 3 cases. Korean J Pain. 2011 Dec;24(4):239-41. doi: 10.3344/kjp.2011.24.4.239. Epub 2011 Nov 30. No abstract available. PMID 22220248
- [Background] Kukkonen J, Kauko T, Vahlberg T, Joukainen A, Aarimaa V. Investigating minimal clinically important difference for Constant score in patients undergoing rotator cuff surgery. J Shoulder Elbow Surg. 2013 Dec;22(12):1650-5. doi: 10.1016/j.jse.2013.05.002. Epub 2013 Jul 12. PMID 23850308
- [Background] Gofeld M, Restrepo-Garces CE, Theodore BR, Faclier G. Pulsed radiofrequency of suprascapular nerve for chronic shoulder pain: a randomized double-blind active placebo-controlled study. Pain Pract. 2013 Feb;13(2):96-103. doi: 10.1111/j.1533-2500.2012.00560.x. Epub 2012 May 4. PMID 22554345
- [Background] Chester R, Shepstone L, Daniell H, Sweeting D, Lewis J, Jerosch-Herold C. Predicting response to physiotherapy treatment for musculoskeletal shoulder pain: a systematic review. BMC Musculoskelet Disord. 2013 Jul 8;14:203. doi: 10.1186/1471-2474-14-203. PMID 23834747
- [Background] Kuijpers T, van der Windt DAWM, van der Heijden GJMG, Bouter LM. Systematic review of prognostic cohort studies on shoulder disorders. Pain. 2004 Jun;109(3):420-431. doi: 10.1016/j.pain.2004.02.017. PMID 15157703
- [Background] Roach KE, Budiman-Mak E, Songsiridej N, Lertratanakul Y. Development of a shoulder pain and disability index. Arthritis Care Res. 1991 Dec;4(4):143-9. PMID 11188601
- [Background] MacDermid JC, Solomon P, Prkachin K. The Shoulder Pain and Disability Index demonstrates factor, construct and longitudinal validity. BMC Musculoskelet Disord. 2006 Feb 10;7:12. doi: 10.1186/1471-2474-7-12. PMID 16472394
- [Background] Roy JS, MacDermid JC, Woodhouse LJ. Measuring shoulder function: a systematic review of four questionnaires. Arthritis Rheum. 2009 May 15;61(5):623-32. doi: 10.1002/art.24396. PMID 19405008
- [Background] Sintonen H. The 15D instrument of health-related quality of life: properties and applications. Ann Med. 2001 Jul;33(5):328-36. doi: 10.3109/07853890109002086. PMID 11491191
- [Background] Vartiainen P, Heiskanen T, Sintonen H, Roine RP, Kalso E. Health-related quality of life and burden of disease in chronic pain measured with the 15D instrument. Pain. 2016 Oct;157(10):2269-2276. doi: 10.1097/j.pain.0000000000000641. PMID 27355183
- [Background] Kane TP, Rogers P, Hazelgrove J, Wimsey S, Harper GD. Pulsed radiofrequency applied to the suprascapular nerve in painful cuff tear arthropathy. J Shoulder Elbow Surg. 2008 May-Jun;17(3):436-40. doi: 10.1016/j.jse.2007.10.007. Epub 2008 Mar 7. PMID 18328740
- [Background] Gurbet A, Turker G, Bozkurt M, Keskin E, Uckunkaya N, Sahin S. [Efficacy of pulsed mode radiofrequency lesioning of the suprascapular nerve in chronic shoulder pain secondary to rotator cuff rupture]. Agri. 2005 Jul;17(3):48-52. Turkish. PMID 16158343